CLINICAL TRIAL: NCT02022371
Title: Prostate Cancer Genomic Heterogeneity
Acronym: PROGENY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Hashim Uddin Ahmed, MRC Clinician Scientist, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13/0244
Record Dates: First submitted 2013-12-15; First posted 2013-12-27 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: PROSTATE CANCER
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Targeted biopsy (Experimental): Snap frozen targeted biopsies of the prostate for genomic analysis
  Interventions: Procedure: Targeted biopsies of the prostate

INTERVENTIONS:
Procedure: Targeted biopsies of the prostate — Multiple biopsies from a MRI lesion for analysis of intratumour heterogeneity
  Other Names: SmartTarget Biopsies of the prostate for snap frozen tissue in order to obtain genetic heterogeneity

SUMMARY:
The purpose of this study is to carry out very detailed genetic testing on prostate cancer cells. The reason to do this is because researchers do not fully understand

* How prostate cancer develops
* Why some cancer cells spread and others do not
* Why some cancer cells respond to treatment and others do not

Researchers and doctors know that 1 in 3 of the male population over the age of 50 has cancer cells in their prostate. However, most of these men will never know they have it and it will not affect their quality of life or their life expectancy. However, some cancers can be aggressive. These are more likely to spread outside of the prostate and cause problems. Doctors do not have an accurate way to tell the difference between aggressive cancer and those which will not cause any problems. Even within one prostate some tumours are aggressive and others do not cause a problem during the lifetime of a patient. In fact, even within one tumour, different cells may behave differently. In other words, one part of the tumour may be aggressive and spread, whilst another part of the same tumour does not. This project will try to find out more about what makes different tumours and different parts of the same tumour aggressive or harmless.

It is important to find out what makes some cancer cells spread and others stay where they are. For the investigators to do this they need to collect fresh samples of cancer tissue from the prostate and from different areas of a tumour within the prostate. This is because biopsies used to diagnose or exclude cancer by the hospital laboratory are not good enough to give investigators detailed genetic information. These biopsies have been put into a chemical called formalin which reduces the quality of the genetic information.

Investigators are therefore asking patients who are undergoing prostate biopsies as part of their normal care to allow them to take additional biopsies for the purpose of this study. This may be the first time patients are having biopsies. Or, patients may be having biopsies after treatment that has been given for the cancer and the doctors are concerned the treatment is not working.

DETAILED DESCRIPTION:
Cancer is a genetic disease, caused by mutations in genes that lead to increased cell proliferation and survival. Importantly, the genetic changes vary dramatically between individual prostate cancer patients and the specific combination of mutations within a patient's cancer is thought to determine tumour aggressiveness and clinical outcome.

Personalized medicine approaches aim to decipher the genetic code of a patient's tumour in order to identify cancers which will behave aggressively and need treatment. However, extensive intra-tumour heterogeneity (ITH) has been discovered in several solid tumour types, complicating the identification of the relevant genetic changes as they may not be present throughout the entire tumour and are likely to be missed by tumour biopsies. ITH is thus a major hurdle for the implementation of personalized cancer treatment approaches.

Investigators have developed genetic technologies that allow them to measure ITH in solid tumours and they now want to apply these to patients with prostate cancer to define the extent and the clinical importance of ITH in this disease which is currently unknown. This will involve looking at the control of genes in the cancer cells which make some tumours more aggressive than others. This may help in predicting which tumours are important and need to be targeted and those that could be left so that too much tissue damage does not occur as a result of therapy. Finding out why some cancer cells spread and others do not may also help to identify novel molecular targets that could be used to prevent the development of metastases.

Patients with suspected prostate cancer usually have scans and then prostate biopsies. These biopsies are needed by the pathologist to make a proper diagnosis and cannot be used for full genetic analysis. So, investigators will ask patients whether they would be willing to give some extra samples of tissue while undergoing these routine biopsies.

Defining ITH in prostate cancer will provide important insights into the genetics of prostate cancer development and metastatic progression and is a key prerequisite for the development of reliable personalized cancer medicine approaches. Thus this study will significantly advance researchers' efforts to predict which tumours are dangerous and in need of urgent treatment and those that could safely be left untreated which would spare these patients the unnecessary side effects. Investigators think that this research work will have a major impact on the use of next generation sequencing in the management of prostate cancer through an in-depth understanding of how common are differences between and within individual cancer lesions. Investigators also want to find out whether these differences, if they exist, are important in tumour development and spread to other areas. Investigators think that the characterization of these differences will allow them to successfully use this information to group patients undergoing treatment using molecular 'signatures' so that treatment is targeted rather than applied in a 'sledge-hammer' approach. Investigators believe that without studies like PROGENY, doctors will instead rely on data from single tumour biopsies which can be misleading since single biopsies may not have sampled the most aggressive tumour area. Finally, investigators think that PROGENY will reveal how prostate cancers evolve over time and which of these changes lead to metastases and ultimately kill the patient. These are called phylogenetic studies and will help work out the main (or 'trunk') genomic changes from later events in 'branches'. This may allow researchers to focus their drug discovery efforts on the common 'trunk' genomic changes.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve group

  1. Men with no prior diagnosis of prostate cancer undergoing prostate biopsy based on identified lesions on imaging
  2. Men with a raised PSA above 15ng/ml
  3. Men giving informed consent

Treated men

1. Men undergoing tissue biopsy for suspicion of prostate cancer recurrence following previous local or systemic therapy based on identified lesions in multi-parametric MRI, bone-scan, choline PET/CT, or PET/MRI

   Exclusion Criteria:
   * 1. Unable to have MRI scan or CT scan, or in whom artefact would reduce scan quality
2. Unable to have prostate biopsy
3. Unable to undergo biopsy for metastatic evaluation
4. On immunosuppression or predefined immunosuppressed state
5. A coagulopathy predisposing to bleeding
6. Unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Tumour heterogeneity | At time of biopsy
  To define the extent of inter/intra-tumour heterogeneity and its association with disease stage at diagnosis and Gleason grade by deep genomic sequencing of multiple regions of intermediate Gleason grade tumours and high Gleason grade tumours, with and without metastatic disease.
Clonal origin of secondary tumours | At time of biopsy
  Through clonal re-ordering and multi-regional prostate mapping, determine whether satellite tumour nodules in high grade prostate cancers represent monoclonal disease related to the index lesion or the evolution of polyclonal cancers by evaluating the deep genomic signatures of primary and secondary lesions within the prostate
Relationship of tumours to metastases | At time of biopsy
  Identify genotype requirements for metastasis development by deep sequencing DNA from the associated metastases from the same patient to reconstruct clonal evolution from primary tumour to metastatic sites and identify evolutionary bottlenecks governing metastasis development that may be targetable for clinical benefit.

SECONDARY OUTCOMES:
Identifying genomic signature of tumour DNA in blood | At time of biopsy
  To determine whether ultra-deep sequencing of circulating plasma DNA can reconstruct inter/intra-tumour heterogeneity and clonal evolution occurring in men who have failed first- and second-line therapies (for localized and metastatic disease).
Genomic signature changes in tumour DNA in blood when drug resistance develops | At time of biopsy
  To determine whether ultra-deep sequencing of circulating plasma DNA can reconstruct inter/intra-tumour heterogeneity and clonal evolution occurring during the acquisition of castration resistant disease.
Relationship of tumour genomics with imaging | At time of biopsy
  To determine the association of inter/intra-tumour heterogeneity with functional imaging with multi-parametric magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals, London, United Kingdom

REFERENCES:
- [Derived] Linch M, Goh G, Hiley C, Shanmugabavan Y, McGranahan N, Rowan A, Wong YNS, King H, Furness A, Freeman A, Linares J, Akarca A, Herrero J, Rosenthal R, Harder N, Schmidt G, Wilson GA, Birkbak NJ, Mitter R, Dentro S, Cathcart P, Arya M, Johnston E, Scott R, Hung M, Emberton M, Attard G, Szallasi Z, Punwani S, Quezada SA, Marafioti T, Gerlinger M, Ahmed HU, Swanton C. Intratumoural evolutionary landscape of high-risk prostate cancer: the PROGENY study of genomic and immune parameters. Ann Oncol. 2017 Oct 1;28(10):2472-2480. doi: 10.1093/annonc/mdx355. PMID 28961847